CLINICAL TRIAL: NCT06516978
Title: A Prospective, Open-Label, Multicenter, Randomized Controlled Study Comparing the Efficacy and Safety of Polatuzumab Vedotin, Rituximab, Cyclophosphamide, Doxorubicin, and Prednisone Combined With Orelabrutinib/Chidamide/Venetoclax/Lenalidomide/PD1 (Pola-RCHP-X) Versus RCHOP-X and Pola-RCHP in Previously Untreated Patients With Diffuse Large B-Cell Lymphoma
Brief Title: A Study Comparing the Efficacy and Safety of Pola-RCHP-X Versus RCHOP-X and Pola-RCHP in Previously Untreated Patients With DLBCL
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, WEI XU, M.D, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-SR-436
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — polatuzumab vedotin; Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; orelabrutinib; venetoclax; N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; penpulimab; Lenalidomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Pola-RCHP-X (Experimental): From cycles 1 to 6, patients will receive Polatuzumab Vedotin 1.8 mg/kg, Rituximab 375 mg/m², Cyclophosphamide 750 mg/m², and Doxorubicin 50 mg/m² on day 1 of each cycle, and Prednisone 100 mg/day from days 1 to 5. From cycles 2 to 6, patients will receive either Orelabrutinib 150 mg/day (days 1-21), Venetoclax 800 mg (days 4-10 in cycle 2; days 1-10 in cycles 3-6), Chidamide 20 mg/day (days 1, 4, 8, 11), Penpulimab 200 mg/day (day 0), or Lenalidomide 25 mg/day (days 1-10). In cycles 7 to 8, patients will receive Rituximab 375 mg/m² on day 1 of each cycle.
  Interventions: Drug: Polatuzumab vedotin; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Prednisone; Drug: Orelabrutinib; Drug: Venetoclax; Drug: Chidamide; Drug: Penpulimab; Drug: Lenalidomide
- RCHOP-X (Active Comparator): From cycles 1 to 6, patients will receive Rituximab 375 mg/m², Cyclophosphamide 750 mg/m², Doxorubicin 50 mg/m², and Vincristine 1.4 mg/m² on day 1 of each cycle, and Prednisone 100 mg/day from days 1 to 5. From cycles 2 to 6, patients will receive either Orelabrutinib 150 mg/day (days 1-21), Venetoclax 800 mg (days 4-10 in cycle 2; days 1-10 in cycles 3-6), Chidamide 20 mg/day (days 1, 4, 8, 11), Penpulimab 200 mg/day (day 0), or Lenalidomide 25 mg/day (days 1-10). In cycles 7 to 8, patients will receive Rituximab 375 mg/m² on day 1 of each cycle.
  Interventions: Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone; Drug: Orelabrutinib; Drug: Venetoclax; Drug: Chidamide; Drug: Penpulimab; Drug: Lenalidomide
- Pola-RCHP (Active Comparator): From cycles 1 to 6, patients will receive Polatuzumab Vedotin at 1.8 mg/kg, Rituximab at 375 mg/m², Cyclophosphamide at 750 mg/m², and Doxorubicin at 50 mg/m² on day 1 of each cycle, and Prednisone at 100 mg/day from days 1 to 5. In cycles 7 to 8, patients will receive Rituximab at 375 mg/m² on day 1 of each cycle.
  Interventions: Drug: Polatuzumab vedotin; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Prednisone

INTERVENTIONS:
Drug: Polatuzumab vedotin — Polatuzumab vedotin IV infusion will be administered as per the schedule specified in the respective arm.
  Arms: Pola-RCHP; Pola-RCHP-X
Drug: Rituximab — Rituximab IV infusion will be administered as per the schedule specified in the respective arm.
Drug: Cyclophosphamide — Cyclophosphamide IV infusion will be administered as per the schedule specified in the respective arm.
Drug: Doxorubicin — Doxorubicin IV infusion will be administered as per the schedule specified in the respective arm.
Drug: Vincristine — Vincristine IV infusion will be administered as per the schedule specified in the respective arm.
  Arms: RCHOP-X
Drug: Prednisone — Prednisone PO will be administered as per the schedule specified in the respective arm.
Drug: Orelabrutinib — Orelabrutinib PO will be administered as per the schedule specified in the respective arm.
  Arms: Pola-RCHP-X; RCHOP-X
Drug: Venetoclax — Venetoclax PO will be administered as per the schedule specified in the respective arm.
  Arms: Pola-RCHP-X; RCHOP-X
Drug: Chidamide — Chidamide PO will be administered as per the schedule specified in the respective arm.
  Arms: Pola-RCHP-X; RCHOP-X
Drug: Penpulimab — Penpulimab IV infusion will be administered as per the schedule specified in the respective arm.
  Arms: Pola-RCHP-X; RCHOP-X
Drug: Lenalidomide — Lenalidomide PO will be administered as per the schedule specified in the respective arm.
  Arms: Pola-RCHP-X; RCHOP-X

SUMMARY:
This study aims to compare the efficacy and safety of Polatuzumab Vedotin, Rituximab, Cyclophosphamide, Doxorubicin, and Prednisone combined with Orelabrutinib/Chidamide/Venetoclax/Lenalidomide/PD1 (Pola-RCHP-X) versus RCHOP-X and Pola-RCHP in previously untreated patients with DLBCL.

ELIGIBILITY:
Inclusion Criteria:

* Sign the informed consent form
* Previously untreated participants with CD20-positive DLBCL
* Life expectancy ≥ 6 months
* IPI score 2-5
* ECOG Performance Status of 0, 1, or 2
* Left ventricular ejection fraction (LVEF) ≥ 50% on cardiac multiple-gated acquisition (MUGA) scan or cardiac echocardiogram (ECHO)
* Adequate hematologic function (unless due to underlying disease, as established for example, by extensive bone marrow involvement or due to hypersplenism secondary to involvement of the spleen by DLBCL per the investigator for which blood product transfusions are permitted) defined as follows:

Hemoglobin ≥ 9.0 g/dL without packed RBC transfusion during 7 days before first treatment ANC ≥ 1.0 x 10^9/L PLT ≥ 75 x 10^9/L

Exclusion Criteria:

* Contraindication to any of the individual components of Pola-RCHP or Orelabrutinib/Chidamide/Venetoclax/Lenalidomide/PD1
* History of other malignancy that could affect compliance with the protocol or interpretation of results
* Significant or extensive history of cardiovascular disease such as New York Heart Association Class III or IV cardiac disease or Objective Assessment Class C or D, myocardial infarction within the last 6 months prior to the start of Cycle 1, unstable arrhythmias, or unstable angina
* History or presence of an abnormal ECG that is clinically significant in the investigator's opinion
* Any active infection within 7 days prior to Cycle 1 Day 1 that would impact participant safety
* Any of the following abnormal laboratory values (unless any of these abnormalities are due to underlying lymphoma):

Serum AST and ALT ≥ 2.5 x ULN Total bilirubin ≥ 1.5 x ULN Serum creatinine clearance < 40 mL/min (using Cockcroft-Gault formula)

* Suspected active or latent tuberculosis (as confirmed by a positive interferon-gamma release assay)
* Participants with a history of progressive multifocal leukoencephalopathy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 528 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2028-10-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival at 24 months (PFS24) Assessed by Investigator per Lugano Response Criteria for Malignant Lymphoma | At 24 months

SECONDARY OUTCOMES:
Complete Response Rate (CRR) Assessed by Investigator per Lugano Response Criteria for Malignant Lymphoma | End of treatment visit (6-8 weeks after last dose on Day 1 of Cycle 8 [Cycle length=21 days]
Overall Response Rate (ORR) Assessed by Investigator per Lugano Response Criteria for Malignant Lymphoma | End of treatment visit (6-8 weeks after last dose on Day 1 of Cycle 8 [Cycle length=21 days]
Event Free Survival (EFS) Assessed by Investigator per Lugano Response Criteria for Malignant Lymphoma | up to approximately 48 months
Overall Survival (OS) | up to approximately 48 months
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | From enrollment to study completion, a maximum of 48 months